CLINICAL TRIAL: NCT04322227
Title: Interventional, Randomized, Double-blind, Placebo-controlled Three-way Crossover Study Investigating the Pharmacodynamic Effects of Two Doses of Foliglurax Using Electroencephalography in Patients With Parkinson's Disease and in Healthy Subjects
Brief Title: Study Investigating Effects of Foliglurax in Patients With Parkinson's Disease (PD) and Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study termination due to efficacy results of another study
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 18240A
Record Dates: First submitted 2020-01-29; First posted 2020-03-26 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Parkinson Disease; Healthy
MeSH Terms: conditions — Parkinson Disease | interventions — foliglurax

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy (Experimental)
  Interventions: Drug: Foliglurax 10 mg (treatment A); Drug: Foliglurax 30 mg (treatment B); Drug: Placebo (treatment C)
- PD (Experimental)
  Interventions: Drug: Foliglurax 10 mg (treatment A); Drug: Foliglurax 30 mg (treatment B); Drug: Placebo (treatment C)

INTERVENTIONS:
Drug: Foliglurax 10 mg (treatment A) — Foliglurax 10 mg, (BID) capsules, orally
Drug: Foliglurax 30 mg (treatment B) — Foliglurax 30 mg, BID capsules, orally
Drug: Placebo (treatment C) — Placebo, BID capsules, orally

SUMMARY:
The purpose of this study is to investigate effects of foliglurax on brain wave patterns (electric signals) in healthy subjects and in patients with PD

DETAILED DESCRIPTION:
All Treatment Periods (P1 to P3) consist of 7 days of dosing (D1 to D7) with either:

* 10 mg foliglurax bis in die (BID) (treatment A)
* 30 mg foliglurax BID (treatment B)
* Placebo BID (treatment C)

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects

* The subject has an acceptable resting EEG at the Screening Visit, as judged by the investigator
* The subject is, in the opinion of the investigator, generally healthy based on the assessment of medical history, physical examination, vital signs, body weight, ECG, and the results of the haematology, clinical chemistry, urinalysis, serology, and other laboratory tests.

Patients with PD

* The patient has an acceptable resting EEG performed at the screening period, as judged by the investigator.
* The patient is, in the opinion of the investigator, fit for enrolment in the study based on the assessment of medical history, physical examination, vital signs, body weight, ECG, and the results of the haematology, clinical chemistry, urinalysis, serology, and other laboratory tests.
* The patient has been diagnosed with idiopathic PD for ≥3 years, with a current disease severity of 2 to 4 on the modified Hoehn and Yahr scale in the 'off' state.
* The patient has dyskinesia that is not too severe to cause discomfort for the patient during the EEG assessments

Exclusion criteria:

* The subject has taken disallowed medication <1 week prior to the first dose of Investigational Medicinal Product (IMP) or <5 half-lives prior to the Screening Visit for any medication taken.
* The subject has significant alcohol consumption
* The subject has taken any investigational medicinal product <3 months prior to the first dose of IMP.
* The subjects has a known genetic disorder of human UDPglucoronosyltransferase
* The subject is pregnant or breastfeeding.

Other in- and exclusion criteria may apply

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Latency of EEG movement related desynchronization of the μ-oscillations | From baseline to Day 7 in each Treatment Period
  Latency of μ-desynchronization ipsilateral and contralateral (in ms)
Latency of EEG movement related synchronization of the beta-oscillations | From baseline to Day 7 in each Treatment Period
  Latency of beta-rebound ipsilateral and contralateral (in ms)
Offset of EEG movement related synchronization of the beta-oscillations | From baseline to Day 7 in each Treatment Period
  Offset of beta-rebound ipsilateral and contralateral (in ms)
Latency of movement from cue measured by accelerometer | From baseline to Day 7 in each Treatment Period
  Latency of movement from cue (in ms)
Average power in u-desynchronization cluster measured by EEG | From baseline to Day 7 in each Treatment Period
  Power in μ-desynchronization cluster ipsilateral and contralateral (in micro-volts squared)
Average power in beta-rebound cluster measured by EEG | From baseline to Day 7 in each Treatment Period
  Power in beta-rebound cluster ipsilateral and contralateral (in micro-volts squared)
Power in the frequency domain of the greater tremor frequency | From baseline to Day 7 in each Treatment Period
  Power in micro-volts squared

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- Biotrial Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: Undecided